CLINICAL TRIAL: NCT06926166
Title: Human Genes and Microbiota in Early Life (HuGME)
Brief Title: Human Genes and Microbiota in Early Life
Acronym: HuGME
Status: Recruiting | Type: Observational
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Principal Investigator, Xiu Qiu, The division of the born in Guangzhou cohort study, Guangzhou Women and Children's Medical Center
Other Study IDs: 201807010086; 82003471 (Other Grant/Funding Number: National natural science foundation of China); 2021A1515110194 (Other Grant/Funding Number: GuangDong Basic and Applied Basic Research Foundation); SL2024A04J0217 (Other Grant/Funding Number: Guangzhou Science and Technology Project)
Record Dates: First submitted 2025-03-26; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Host and Microbiome; Pregnancy Outcomes; Pregnancy Complications; Neurodevelopmental Disorders; Immune Development; Childhood Obesity; Type 2 Diabetes
MeSH Terms: conditions — Pregnancy Complications; Neurodevelopmental Disorders; Pediatric Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — During pregnancy: maternal blood, urine, and stool. At delivery: cord, cord blood, and placenta. During infancy: dry blood spots, stool, and blood. During childhood: blood, buccal swab, and stool.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- No treatment: No treatment
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The long-term goal of the Human Genes and Microbiota in Early Life (HuGME) is to explore the short- and long-term effects of maternal microbiota during pregnancy and the microbiota colonization of their offspring early in life and their interaction with the host on maternal-offspring health consequences in later life in the born in Guangzhou cohort study in China. Identification of the effect of microbiota in early life, as well as environmental factors and microbe-host interaction, will lead to a better understanding of disease pathogenesis and provide a foundation for targeted mechanistic investigation into the consequences of microbial-host crosstalk for long-term health. It also can result in new strategies to predict and prevent diseases in later life.

DETAILED DESCRIPTION:
Prenatal and early postnatal life represent critical windows for growth and cognitive and immune system development. In addition to genetics and host biology, the environment plays a critical role in the health of a child. One key player in this process is the maternal and infant gut microbiomes. The establishment and progression of the intestinal microbiota from birth to childhood are dependent on a range of factors, including maternal microbiota, diet, environment, and medical exposures. The host-microbial crosstalk during this time is thought to be involved in the pathobiology of later-life diseases, such as allergic disease, obesity, and neurodevelopmental delay. Although the microbiome and its importance for health have been extensively studied, it remains unclear how maternal microbiota-fetal interaction, the establishment, and progression of microbiota in infant adaptation to postnatal environmental exposures, and microbial-host crosstalk affect the health of the children in later life.

Hypotheses:

1. Maternal microbiota-fetal interaction has an essential effect on fetal immune system development and adverse pregnancy outcomes.
2. Host genes can shape infant gut microbial assembly and metabolism.
3. Early-life interactions between host genes and microbiota have an impact on immune system development and atopic disease in later life.
4. Co-metabolism of the gut microbiome and metabolites in the host affects childhood obesity
5. Early-life interactions between the host and microbiota have an impact on the neurodevelopment of the children.
6. Maternal microbiota influence the metabolism of the mother during pregnancy and postpartum.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women with < 20 weeks of gestation Pregnant women intended to eventually deliver in Guangzhou Women and Children's medical center Permanent residengts of families intended to remain in Guangzhou with their child for ≥3 years

Exclusion Criteria:

Refuses to have blood and stool samples stored at Born in Guangzhou cohort study Biobank.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women attending their first routine antenatal examinations (usually around week 16) and their partners and offsrping
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2038-12-31 (Estimated); Study Completion 2038-12-31 (Estimated)

PRIMARY OUTCOMES:
Numbers of participants with Childhood diseases. Including: | 42 days, 6 months, 1, 3, 6, 8-9, 14, and18 years of age
  Obesity，asthma，allergic diseases，Delayed neural development，type 1 diabetes，maturity-onset diabetes of the young（MODY), hypertension
Numbers of participants with maternal diseases. Including: | during pregnancy, 42 days, 6 months, 1, 3, 6, 8-9, 14, and18 years after delivery
  Obesity，asthma，allergic diseases，type 1 diabetes，type 2 diabetes, hypertension , cardiovascular diseases，and obstetric complications，including gestational diabetes，pregnancy induced hypertension, ect.

SECONDARY OUTCOMES:
Neurodevelopment during early childhood | at age of 3 years
  Including adaptive, gross motor, fine motor,language,and social function; assessed using Gesell Developmental Schedules
Neurodevelopment during early childhood | at age of 3 years
  Including adaptive, gross motor, fine motor,language,and social function; assessed using Ages and Stages Questionnaire
Neurodevelopment during preschool age | at age of 6 years
  Including solving skills, pattern perception, and logical thinking；assessed using Raven's Standard Progressive Matrices
Neurodevelopment during preschool age | at age of 6 years
  Including solving skills, pattern perception, and logical thinking；assessed using Peabody Picture Vocabulary Test
Neurodevelopment during preadolescence | at age of 8-9 years
  Including higher-level cognitive processes such as attention, perseverance, WM, abstract thinking, CF, and set shifting;assessed using Raven's Standard Progressive Matrices
Neurodevelopment during preadolescence | at age of 8-9 years
  Including higher-level cognitive processes such as attention, perseverance, WM, abstract thinking, CF, and set shifting;assessed using Wsiconsin card sorting test
maternal and childhood abnormal glucose metabolism after delivery | 3, 6 and 9 years after delivery
  blood glucose level：glycosylated hemoglobin，fasting blood glucose, 1-hour glucose, 2-hour glucose, ect.
maternal and childhood abnormal lipid metabolism after delivery | 3, 6 and 9 years after delivery
  Lipid level : total cholesterol, triglycerides, LDL, HDL, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Xiu Qiu, PhD, Principal Investigator — Study Principal Investigator Guangzhou Women and Children's Medical Center, China
Locations (1):
- Guangzhou Women and Children's Medical Center, China, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Qiu X, Lu JH, He JR, Lam KH, Shen SY, Guo Y, Kuang YS, Yuan MY, Qiu L, Chen NN, Lu MS, Li WD, Xing YF, Zhou FJ, Bartington S, Cheng KK, Xia HM. The Born in Guangzhou Cohort Study (BIGCS). Eur J Epidemiol. 2017 Apr;32(4):337-346. doi: 10.1007/s10654-017-0239-x. Epub 2017 Mar 20. PMID 28321694
- [Background] Kuang YS, Lu JH, Li SH, Li JH, Yuan MY, He JR, Chen NN, Xiao WQ, Shen SY, Qiu L, Wu YF, Hu CY, Wu YY, Li WD, Chen QZ, Deng HW, Papasian CJ, Xia HM, Qiu X. Connections between the human gut microbiome and gestational diabetes mellitus. Gigascience. 2017 Aug 1;6(8):1-12. doi: 10.1093/gigascience/gix058. PMID 28873967
- [Background] Gao C, Shao DT, Wang CR, Kuang YS, Lu JH, Zeng DY, He JR, Qiu X. Long-term effect of caesarean section on the gut microbial taxonomical profile and metabolic function of children at pre-school age. Clin Transl Med. 2023 Nov;13(11):e1470. doi: 10.1002/ctm2.1470. No abstract available. PMID 37929652
- [Background] Kuang YS, Li SH, Guo Y, Lu JH, He JR, Luo BJ, Jiang FJ, Shen H, Papasian CJ, Pang H, Xia HM, Deng HW, Qiu X. Composition of gut microbiota in infants in China and global comparison. Sci Rep. 2016 Nov 9;6:36666. doi: 10.1038/srep36666. PMID 27827448
- [Background] Guo Y, Li SH, Kuang YS, He JR, Lu JH, Luo BJ, Jiang FJ, Liu YZ, Papasian CJ, Xia HM, Deng HW, Qiu X. Effect of short-term room temperature storage on the microbial community in infant fecal samples. Sci Rep. 2016 May 26;6:26648. doi: 10.1038/srep26648. PMID 27226242